CLINICAL TRIAL: NCT06831929
Title: Human Papillomavirus Ends Here: A Multilevel Intervention to Increase Uptake of the HPV Vaccine Among Adolescents
Brief Title: HPV Ends Here: Increasing Uptake of the HPV Vaccine
Acronym: HPV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2179292-1; 1K01CA258956-01A1 (NIH)
Record Dates: First submitted 2025-02-06; First posted 2025-02-18 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: HPV Vaccine
Keywords: HPV; Human Papillomavirus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (No Intervention): These clinics will not receive any intervention and will continue with care as usual.
- Intervention Arm (Experimental): These clinics will receive the multilevel intervention which will include tailored parent/patient education, appointment scheduling assistance, and primary care team trainings.
  Interventions: Behavioral: Intervention Arm

INTERVENTIONS:
Behavioral: Intervention Arm — Within the intervention clinics, parents of patients between the ages of 10-12 (who are eligible for the HPV vaccine) will receive a culturally tailored customized HPV vaccine message and testimonial video from a patient/survivor of an HPV associated cancer (e.g., oropharyngeal, or cervical) via the MyChart patient portal. Parents will also receive a personal call from the research coordinator to remind them that their child is due for the HPV vaccine. If the parent is interested in scheduling the HPV vaccine appointment during this call, the research coordinator will transfer the parent to UC Davis appointment call center to schedule the appointment. Also, primary care team members will receive a semi-annual learn at lunch workshop focused on strategies to introduce the HPV vaccine to parents and how to address concerns from vaccine hesitant parents. Workshop content will be tailored/adapted to include patient/parent cultural considerations.
  Arms: Intervention Arm

SUMMARY:
Develop, implement, and evaluate a culturally tailored multilevel intervention to increase uptake of the HPV vaccine among eligible patients ages 10-12 of the University of California, Davis Health Community Physician (UCDH CP) primary care practices using a randomized controlled trial design.

DETAILED DESCRIPTION:
The goal of this study is to use an evidence-based approach to develop, implement and evaluate a ML intervention on increasing HPV vaccine uptake among UCDH CP patients ages 10-12.

Aim 1. Refine and finalize a parent, primary care team and clinic ML intervention to increase uptake and completion of the HPV vaccine series among adolescent patients of the UCDH CP practices. In Phase 1, semi-structured qualitative interviews with key stakeholders will be conducted to refine the content and implementation approaches.

Aim 2. Conduct and evaluate the effectiveness and sustainability of the ML intervention. In Phase 2, twelve UCDH CP practices will be recruited to participate in a 2-arm parallel group randomized controlled trial. The primary outcome age-appropriate completion of the HPV vaccine series will be assessed via Epic, the UCDHS electronic medical record (EMR) software. It is hypothesized that patients of clinics in the intervention condition will have significantly higher HPV completion rates compared to patients of clinics in the control condition (usual care).

ELIGIBILITY:
Inclusion Criteria:

• Clinic patients between the ages of 10-12 who are eligible for the HPV vaccine

Exclusion Criteria:

• Clinic patients who already received the HPV vaccine or with any contraindication to the HPV vaccine.

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2232 (Estimated)
Dates: Start 2025-02-28 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome: Evaluation | One year
  Number of participants who initiate and complete the HPV vaccine series

CONTACTS AND LOCATIONS:
Overall Officials: Julie HT Dang, PhD, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Health, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No